CLINICAL TRIAL: NCT01480752
Title: the Effect of Intraligamentary Injection of Lornoxicam on the Intensity of Post-operative Endodontic Pain in the Tooth With Symptomatic Irreversible Pulpitis
Brief Title: Reduction of Post-operative Endodontic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Mandana Abedi Tari, principal investigator, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRCT201108017191N1
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Post Operative Endodontic Pain
Keywords: In the patients with symptomatic Irreversible Pulpitis
MeSH Terms: interventions — lornoxicam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lornoxicam (Active Comparator)
  Interventions: Drug: Lornoxicam
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline
- no injection (Placebo Comparator)
  Interventions: Drug: no injection

INTERVENTIONS:
Drug: Lornoxicam — PDL injection of 0/2 ml of lornoxicam (4mg/ml),before the root therapy and after the inferior alveolar injection
  Other Names: Xefo; (904111)
  Arms: Lornoxicam
Drug: normal saline — PDl injection of 0/2 ml normal saline before the root therapy and after inferior alveolar injection
  Arms: normal saline
Drug: no injection — inject nothing after inferior alveolar injection and before root canal therapy
  Arms: no injection

SUMMARY:
To determine the effect of intraligamentary injection of Lornoxicam on the intensity of post-operative endodontic pain in the tooth with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
sixty qualified samples (initial estimate which will be come more accurate after the pilot study on 6 patients) will be divided randomly in three groups which all of them will have an inferior Alveolar injection and before the beginning of the treatment the primary group will receive an injection of 0.4 mL ( 0.2 mL in mesio buccal and 0.2 mL in disto buccal) of Lornoxicam and the second group will be injected with 0.4 mL of normal saline( 0.2 mL in mesio buccal and 0.2 mL in disto buccal) ,in third group we will only pretend the injection but actually there is no substance injected ,making the patient believe that there was an injection . Then the patients' pain will be evaluated with visual Analogue Scale analysis (VAS) 0-170 mm in time intervals of 6, 12, 24 and 48 hours after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* healthy (ASA I, II);
* Patients with first or second mandibular molars who need endodontic treatment;
* Vital tooth without a history of past endodontic treatment;
* Patients with clinical evidence of irreversible Pulpits with moderate to severe pain;
* Patients without pre apical lesion and periodontal ligament enlargement more than 0.75-1mm on the x-ray images;
* Patients in the age group of 18-65 years old

Exclusion Criteria:

* Pregnant or nursing;
* necrotic tooth;
* Patients with allergy or contraindication toward non-opioid or opioid painkillers such as aspirin or NSAIDs;
* People who have a history of acute peptic ulcer, during the past 12 months;
* People who have bleeding problems or have been taking anticoagulant drugs over the past month;
* Patients who have taken opioid or non opioid or steroid pain killers, antidepressants or sedative drugs.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Post operative endodontic's pain | 6,12,24,48 hours after drug's injection
  The measuring method of the pain is VAS(Visual Analogue Scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Dental School of Azad University, Tehran, Tehran Province, Iran